CLINICAL TRIAL: NCT01560403
Title: A One-Year, Open-Label Study With Teduglutide for Subjects With Parenteral Nutrition-dependent Short Bowel Syndrome Who Completed Study CL0600-021
Brief Title: A One-Year, Open-Label Study With Teduglutide for Subjects Who Completed Study CL0600-021
Acronym: STEPS3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED-C11-001
Record Dates: First submitted 2012-03-13; First posted 2012-03-22 (Estimated); Results first posted 2014-12-25 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Short Bowel Syndrome
Keywords: Parenteral nutrition; TPN; HPN; PN; SBS; Short bowel syndrome
MeSH Terms: conditions — Short Bowel Syndrome; Hyperphagia | interventions — teduglutide; ALX-0600

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Teduglutide (Experimental): 0.05 mg/kg/day
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — 0.05 mg/kg/day subcutaneously taken once per day for 12 months
  Other Names: Gattex

SUMMARY:
This study is a 1-year open label extension study to collect long term efficacy and safety data from patients who have completed approximately 2 years of dosing in Study CL0600-021.

DETAILED DESCRIPTION:
This study served as a 1-year extension study for those US patients who have completed the CL0600-021 study.

ELIGIBILITY:
Inclusion Criteria:

* At completion of Study CL0600-021, subjects will be invited to participate in this trial if they meet the following criteria:

  1. Completion of the 24-month study, CL0600-021, regardless if fully weaned from PN/I.V. support
  2. Signed and dated informed consent form (ICF) to participate before any study-related procedures of Study TED-C11-001 are performed

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2013-07-23 (Actual); Study Completion 2013-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (5):
  - Scripps Clinic & Research Foundation, La Jolla, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Mount Sinai Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Result] Seidner DL, Fujioka K, Boullata JI, Iyer K, Lee HM, Ziegler TR. Reduction of Parenteral Nutrition and Hydration Support and Safety With Long-Term Teduglutide Treatment in Patients With Short Bowel Syndrome-Associated Intestinal Failure: STEPS-3 Study. Nutr Clin Pract. 2018 Aug;33(4):520-527. doi: 10.1002/ncp.10092. Epub 2018 May 15. PMID 29761915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 1-year, open-label, multi-center study in subjects who completed Study CL0600-021 (NCT00930644) at any US site.
Groups:
- TED/TED: This group represents those subjects exposed to active treatment with teduglutide for 24 weeks in Study CL0600-020 (NCT00798967) and an additional 24 months in Study CL0600-021 (NCT00930644)
- NT/PBO,TED: This group represents those subjects who either participated in Study CL0600-020 and received placebo, or who were eligible for randomization in Study CL0600-020 (NCT00798967), but qualified after the enrollment number was already satisfied and therefore entered the open-label extension Study CL0600-021 (NCT00930644) directly
Period: Overall Study
Arm/Group | TED/TED | NT/PBO,TED
Started | 5 | 9
Completed | 5 | 8
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- TED/TED: This group represents those subjects exposed to active treatment with teduglutide for 24 weeks in Study CL0600-020 (NCT00798967) and an additional 24 months in Study CL0600 021 (NCT00930644)
- Total: Total of all reporting groups
Arm/Group | TED/TED | NT/PBO,TED | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Customized [Count of Participants; unit: Participants] — Age at Study CL0600-020 (NCT00798967) Informed Consent (year)
  Participants
    < 45 years | 1 | 2 | 3
    45 - < 65 years | 3 | 6 | 9
    >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Summary of Treatment-emergent Adverse Events
Description: As the primary intent of this study was to collect additional safety data, this outcomes measure will provide a summary of the treatment emergent adverse events. Based on the start date of each subject in this study and the study end date, not all subjects reached 12 months.
Time Frame: 12 months
Population: Safety Population
Measure: Number; unit: participants
Groups:
- NT,PBO/TED: This group represents those subjects who either participated in Study CL0600-020 (NCT00798967) and received placebo, or who were eligible for randomization in Study CL0600-020 (NCT00798967), but qualified after the enrollment number was already satisfied and therefore entered the open-label extension study CL0600-021 (NCT00930644) directly.
Arm/Group | NT,PBO/TED | TED/TED
Number analyzed (Participants) | 9 | 5
participants | 4 | 5

ADVERSE EVENTS:
Time Frame: 1 year, 2 months
Description: Date of Study Initiation (first subject, first visit) 21 May 2012 Date of Study Completion (last subject, last visit) 23 July 2013. Due to the different start dates of each subject in this study, not all subjects completed the 12 month visits by the study completion date as the study was terminated on this date by the sponsor.
Arm/Group | NT/PBO,TED | TED/TED
Serious Adverse Events (participants affected / at risk) | 1/9 | 5/5
Other Adverse Events (participants affected / at risk) | 4/9 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NT/PBO,TED (N=9) | TED/TED (N=5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Central line infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NT/PBO,TED (N=9) | TED/TED (N=5)
Asthenic conditions (General disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anxiety symptoms (Psychiatric disorders) | 1 (1) | 1 (1)
Benign neoplasms gastrointestinal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Catheter sepsis (Infections and infestations) | 0 (0) | 2 (2)
Catheter site related reaction (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Cognition and attention disorders and disturbances (Psychiatric disorders) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hepatic enzyme increased (Investigations) | 1 (3) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (3)

LIMITATIONS AND CAVEATS:
This study provided further long-term safety and efficacy data on the 14 US subjects who enrolled in the CL0600-020 and the CL0600-021 study. Given the small number of subjects in this study, only descriptive statistics were employed and presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No